CLINICAL TRIAL: NCT01192945
Title: Piaza - Non-interventional Study on the Efficacy and Safety of Azacitidin (Vidaza®) in Patients With Myelodysplastic Syndromes (MDS, INT-2 or High Risk), AML (WHO 20-30% Blasts), or CMMoL (10-29% Bone Marrow Blasts Without Myeloproliferative Disorder)
Brief Title: Non-interventional Study With Azacitidin (Vidaza®)
Acronym: Piaza
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-0905
Record Dates: First submitted 2010-07-30; First posted 2010-09-01 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-08

CONDITIONS: MDS; AML; CMMOL
Keywords: Azacitidin; Vidaza; Piaza; myelodysplastic syndrome; MDS; chronic myelomonocytic leukemia; CMML; acute myeloid leukemia; AML; daily routine; concomitant antiemetic therapy; germany; non-interventional study
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this non-interventional study is to collect data on the efficiency and safety of Azacitidin in the routine application.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not eligible for haematopoietic stem cell transplantation, who are at least 18 years old (no age limit to top) and who have one of the following diseases:

  * myelodysplastic syndrome (MDS) with intermediate risk 2 or high risk according to the International Prognostic Scoring System (IPSS)
  * chronic myelomonocytic leukemia (CMML) with 10-29% marrow blasts without myeloproliferative disorder
  * acute myeloid leukemia (AML) with 20-30% blasts and multilineage dysplasia according to classification of the World Health Organisation (WHO).

Exclusion Criteria:

* Contraindication according to the summary of product characteristics of Vidaza®
* Signed patient informed consent form is not available
* Patients with advanced malignant hepatic tumors
* Pregnant or nursing women, men and women (of childbearing age) who are unwilling to apply a reliable method of contraception during and up to three months after treatment with Azacitidine
* Necessary or planned treatment with other systemic cytostatics
* Known medical history of severe decompensatoric cardiac insufficiency
* Medical history of clinically unstable cardiac or pulmonary disease
* Known or suspected hypersensitivity to azacitidine or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are not suitable for transplantation of hematopoietic stem cells and have one of the following diseases: myelodysplastic syndrome (MDS) with intermediate risk 2 or high risk according to the International Prognostic Scoring System (IPSS), chronic myelomonocytic leukemia (CMML) with 10-29% marrow blasts without myeloproliferative disorder, acute myeloid leukemia (AML) with 20-30% blasts and multilineage dysplasia according to classification of the World Health Organisation (WHO).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Progression-free-survival | 2 years after LPI

SECONDARY OUTCOMES:
2 year survival rate | 2 years after LPI
overall survival | 2 years after LPI
overall response rate | 2 years after LPI
time to treatment discontinuation | 2 years after LPI
haematological improvement | 2 years after LPI
relative dosage of azacitidine | 2 years after LPI
liver and kidney functionality | 2 years after LPI
blood transfusion requirements | 2 years after LPI
supportive medication | 2 years after LPI

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Wehmeyer, Dr., Principal Investigator — Hämatologisch-onkologische Gemeinschaftspraxis
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany